CLINICAL TRIAL: NCT02168023
Title: Randomised Controlled Trial Evaluating Dialkylcarbamoyl Chloride (DACC) Impregnated Dressings for the Prevention of Surgical Site Infections in Adult Women Undergoing Caesarean Section.
Brief Title: Study to Evaluate DACC Dressings for the Prevention of Surgical Site Infections in Women Undergoing Caesarean Section.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Paweł Stanirowski, Doctor of Medicine, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DACC-1; KB/127/2014 (Other: Ethics Committee approval number)
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Surgical Site Infection; Infection; Cesarean Section
Keywords: surgical site infection; dialkylcarbamoylchloride impregnated dressing; caesarean section; wound dehiscence
MeSH Terms: conditions — Surgical Wound Infection; Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DACC impregnated dressing (Experimental): Patients undergoing elective or emergency caesarean section with DACC impregnated dressing Sorbact Surgical Dressing ® (ABIGO Medical AB, Sweden) placed over post-caesarean wound after skin closure, the dressing will be removed after the first 48 hours postoperatively
  Interventions: Device: DACC impregnated dressing
- Standard surgical dressing (Active Comparator): Patients undergoing elective or emergency caesarean section with standard surgical dressing placed over post-caesarean wound after skin closure, the dressing will be removed after the first 48 hours postoperatively
  Interventions: Device: Standard surgical dressing

INTERVENTIONS:
Device: DACC impregnated dressing — DACC impregnated dressing Sorbact Surgical Dressing ® (ABIGO Medical AB, Sweden) placed over post-caesarean wound after skin closure, the dressing will be removed after the first 48 hours postoperatively
  Other Names: Sorbact Surgical Dressing ® (ABIGO Medical AB, Sweden)
  Arms: DACC impregnated dressing
Device: Standard surgical dressing — Standard surgical dressing placed over post-caesarean wound after skin closure, the dressing will be removed after the first 48 hours postoperatively
  Arms: Standard surgical dressing

SUMMARY:
Surgical site infections (SSIs) constitute an important medical and socioeconomic problem worldwide. Despite the fact that the risk factors for SSIs were identified and the continuously increasing medical knowledge in the fields of tissue engineering, molecular biology and microbiology facilitated the development of numerous new recommendations and methods for management, in many cases the available options for successful treatment of post-operative wound infections remain limited. Non-treated or inappropriately treated SSIs often lead to necrosis of the surrounding tissues, wound dehiscence, formation of fistulas, or become sites of origin for systemic infections. Patients are exposed to risk of further complications and hospitalization time extends resulting in increased total treatment costs. Treatment prolongation affects also the quality of life and psychosocial functioning of patients with impaired wound healing. Considering the arguments above, appropriate prevention and management of infected post-surgical wounds is currently one of the priorities for the majority of invasive medical disciplines.

Obstetrics constitute a field of medicine in which the issues associated with wound healing are particularly relevant. According to the literature data wound infections occur in approximately 1.8-11.3% of women undergoing caesarean section.

Dialkylcarbamoyl chloride (DACC) is a fatty acid derivative that irreversibly binds microorganisms to the dressing fibres as a result of hydrophobic interaction. As the mechanism of DACC action is solely physical no chemical agents are released into the wound bed and the dressing could be safely used by women during puerperal period.

The purpose of this randomized controlled study is to compare the effect of DACC impregnated dressing and standard surgical dressing in the prevention of SSIs in adult women following caesarean section. This study will also evaluate pre-, peri- and postoperative risk factors of SSIs and analyze health economics of DACC impregnated dressings for prevention of post-cesarean wound infections.

DETAILED DESCRIPTION:
This is a single-blinded randomized controlled trial performed at the Department of Obstetrics and Gynecology of Medical University of Warsaw. The study will involve 518 patients undergoing caesarean section who after giving their informed consent will be randomly divided into two groups: study (n=259) and control group (n=259). The study group will receive DACC impregnated dressing - Sorbact Surgical Dressing ® (ABIGO Medical AB, Sweden) and the control group will receive standard surgical dressing.

In all participants transverse skin incision and low transverse uterine incision will be performed during caesarean section procedure.

All participants will receive prophylactic dose of antibiotics prior to the start of surgery (1g cefazolin intravenously 0-30 minutes before surgery) and wound irrigation with octenidine prior to the subcutaneous tissue closure.

For fascial incision, subcutaneous tissue and skin incision closure continuous antibacterial braided absorbable suture, single monofilament absorbable suture and subcuticular continuous monofilament non-absorbable suture will be used, respectively.

Dressing will be left in place for the first 48 hours post caesarean section unless clinical reason exists to replace it. After the first 48 hours postoperatively all of the dressings will be removed and first wound evaluation will be performed. On post-operative day 3 patients will be discharged and indicated to revisit on post-operative day 7 to remove the skin suture. During this follow-up visit second wound review will be performed for any signs of infection. Third, and final wound assessment will take place on post-operative day 14.

To analyze overall treatment costs patients with SSI will be followed up until the end of treatment, up to 8 weeks post surgery.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* undergoing elective or emergency caesarean section
* transverse skin incision
* low transverse uterine incision
* single and multiple pregnancy
* intravenous administration of 1g cefazolin 0-30 minutes prior to the start of surgery
* irrigation of the wound with octenidine prior to the subcutaneous tissue closure

Exclusion Criteria:

* patients age <18 years
* patients physical or mental incapacity to give informed consent
* skin incision other than transverse
* uterine incision other than low transverse
* patients that did not receive routine prophylactic dose of antibiotics prior to the start of surgery
* patients without irrigation of the wound with octenidine prior to the subcutaneous tissue closure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with surgical site infection | within the first 14 days post surgery
  SSI determined according to Centers for Disease Control and Prevention (CDC) criteria

SECONDARY OUTCOMES:
Percentage of patients with SSI associated wound dehiscence | within the first 8 weeks post surgery
Length of the primary and any secondary hospitalization | Day 0 (day of surgery/ the first day of readmission to hospital) until the date of discharge, up to 8 weeks post surgery
Readmissions to hospital due to SSI following caesarean section | within the first 8 weeks post surgery
Percentage of patients with antibiotic treatment due to SSI following caesarean section | within the first 8 weeks post surgery
Surgeons experience | Day 0 (day of surgery)
  resident, ob/gyn specialist with professional experience <5 years, ob/gyn specialist with professional experience ≥5 years
Length of surgery | Day 0 (day of surgery)
  minutes from skin incision until skin closure
Mode of caesarean section | Day 0 (day of surgery)
  elective or emergency; emergency caesarean section defined as caesarean section performed within 30 minutes from decision
Pathogens responsible for SSI | within the first 8 weeks post surgery
  Wound swab testing to be made in all patients presenting clinical symptoms of surgical site infection
Patients age | Day 0 (day of surgery)
Patients race | Day 0 (day of surgery)
Patients parity | Day 0 (day of surgery)
  primiparous or multiparous
Patients pre-gestational weight | Day 0 (day of surgery)
Patients pre-gestational body mass index | Day 0 (day of surgery)
Patients gestational weight gain | Day 0 (day of surgery)
Percentage of patients with nicotine dependence | Day 0 (day of surgery)
Percentage of patients with gestational diabetes mellitus or pre-gestational diabetes mellitus | Day 0 (day of surgery)
Patients haemoglobin concentration prior to the start of surgery | Day 0 (day of surgery)
Patients haemoglobin concentration after the surgery | 24 hours after surgery
Percentage of patients with surgical intervention due to SSI | within the first 8 weeks post surgery

OTHER OUTCOMES:
Cost of antibiotic treatment due to SSI | Day 0 (the first day of antibiotic treatment) until the last day of treatment, up to 8 weeks post surgery
  Price of antibiotics to be calculated according to manufacturer specifications.
Cost of hospital stay due to SSI | Day 0 (day of SSI diagnosis/ the first day of hospital readmission due to SSI) until the end of treatment and discharge, up to 8 weeks post surgery
  Cost of single hospitalization day to be obtained from hospital financial office.
Cost of nursing care due to SSI | Day 0 (day of SSI diagnosis/ the first day of hospital readmission due to SSI) until the end of treatment and discharge, up to 8 weeks post surgery
  Cost of single day nursing care to be obtained from hospital financial office.
Cost of surgical interventions due to SSI | Day 0 (day of surgery), up to 8 weeks post caesarean section
  Cost of surgical intervention to be approximated using Polish National Health Fund specifications for Diagnosis Related Groups and International Classification of Diseases version 10 (ICD-10) codes.
Cost of ambulatory visits due to SSI | Day 0 (day of SSI diagnosis post-discharge) until the last ambulatory visit, up to 8 weeks post caesarean section
  Cost of ambulatory visit to be approximated using Polish National Health Fund specifications for Diagnosis Related Groups and International Classification of Diseases version 10 (ICD-10) codes.

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Stanirowski, MD, Principal Investigator — Chair and Department of Obstetrics and Gynecology, II Faculty of Medicine, Medical University of Warsaw; Włodzimierz Sawicki, MD, PhD, Study Director — Chair and Department of Obstetrics and Gynecology, II Faculty of Medicine, Medical University of Warsaw
Locations (1):
- Chair and Department of Obstetrics and Gynecology, II Faculty of Medicine, Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

REFERENCES:
- [Background] Falk P, Ivarsson ML. Effect of a DACC dressing on the growth properties and proliferation rate of cultured fibroblasts. J Wound Care. 2012 Jul;21(7):327-8, 330-2. doi: 10.12968/jowc.2012.21.7.327. PMID 22886332
- [Background] Ljungh A, Yanagisawa N, Wadstrom T. Using the principle of hydrophobic interaction to bind and remove wound bacteria. J Wound Care. 2006 Apr;15(4):175-80. doi: 10.12968/jowc.2006.15.4.26901. No abstract available. PMID 16620048
- [Background] Gentili V, Gianesini S, Balboni PG, Menegatti E, Rotola A, Zuolo M, Caselli E, Zamboni P, Di Luca D. Panbacterial real-time PCR to evaluate bacterial burden in chronic wounds treated with Cutimed Sorbact. Eur J Clin Microbiol Infect Dis. 2012 Jul;31(7):1523-9. doi: 10.1007/s10096-011-1473-x. Epub 2011 Nov 19. PMID 22113306
- [Background] Derbyshire A. Innovative solutions to daily challenges. Br J Community Nurs. 2010 Sep;Suppl:S38, S40-5. PMID 20852534
- [Background] Opoien HK, Valbo A, Grinde-Andersen A, Walberg M. Post-cesarean surgical site infections according to CDC standards: rates and risk factors. A prospective cohort study. Acta Obstet Gynecol Scand. 2007;86(9):1097-102. doi: 10.1080/00016340701515225. PMID 17712651
- [Background] Butcher, M. DACC antimicrobial technology: a new paradigm in bioburden management. JWC/BSN supplement:1-20, 2011.